CLINICAL TRIAL: NCT04704570
Title: Investigation of The Effects of Remote Exercise Programs and Preventive Training on Muscle Architecture and Functional Level in Asymptomatic Individuals
Brief Title: Remote Exercise Programs and Preventive Training in Asymptomatic Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Yasemin Özel Aslıyüce, Research Assistant, Physiotherapist, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KA-20110
Record Dates: First submitted 2021-01-08; First posted 2021-01-11 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: Healthy People
Keywords: spinal stabilization exercise; tele-rehabilitation; muscle architecture; functional level
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Treatment Group (Experimental): Remotely Exercises 3 times a week, 8 weeks remotely (with video) spinal stabilization exercises
  Interventions: Other: Exercise
- Control Group (Other): Face to Face Exercises 3 times a week, 8 weeks face to face (in clinic) spinal stabilization exercises
  Interventions: Other: Exercise
- Remotely assessment Group-Face to Face Assessment Group (Other): First, a remote evaluation and then a face to face evaluation will be made.
  Interventions: Other: Remotely and face to face evaluation of Functional Capacity Level
- Face to Face Assessment Group-Remotely assessment Group (Other): First, a facet o face evaluation and then a remote evaluation will be made.
  Interventions: Other: Remotely and face to face evaluation of Functional Capacity Level

INTERVENTIONS:
Other: Exercise — Spinal stabilization exercise
  Arms: Control Group; Treatment Group
Other: Remotely and face to face evaluation of Functional Capacity Level — Quality of life assessment (SF-36), and cognitive assessment ((Montreal Cognitive Assessment Scale (MOCA)) will be administered face to face. Functional capacity assessment tests will be administered both face-to-face and remotely. All participants will be administered both remotely and face-to-face. The order of the remote and face-to-face evaluations will be determined by the closed envelope randomization method. The remote evaluation will be done by video interview method under the direction of the researcher. During the remote evaluation, the necessary equipment for the participant will be prepared in the unit in advance. There will be a 10-30 minute rest interval between each evaluation.This application will only be applied at the beginning of the exercise program.After the 8-week program, only face-to-face evaluation will be made.
  Arms: Face to Face Assessment Group-Remotely assessment Group; Remotely assessment Group-Face to Face Assessment Group

SUMMARY:
In recent years, it has been emphasized that preventive approaches are a less costly and more effective way to treat a pathology. Primary preventive approaches should become widespread, especially in problems with changeable risk factors such as spine health. Various preventive approaches and exercise training seem to be an effective way to prevent the development of back and neck pain. Again, in recent years, the pandemic process has increased the interest and need for tele-rehabilitation. As a result, scientific research results on tele-rehabilitation are needed as a necessity to adapt to the Covid-19 epidemic and the globalizing world. The aim of the thesis study planned in this context is to investigate the effectiveness of remote exercise applications on lumbar and cervical region muscle architecture and functionality in asymptomatic individuals.Another aim of this study is to investigate the remote applicability of functional level, quality of life, kinesophobia and cognitive assessment.

ELIGIBILITY:
Inclusion Criteria:

* Have not experienced back and neck pain for at least 3 months,
* Between the ages of 18-55,
* Literate,
* Individuals who are capable of understanding exercises (Montreal Cognitive Assessment Scale (MOCA) (19) total score> 21) will be included in the study.

Exclusion Criteria:

* Having been diagnosed with cervical or lumbar region pathologies,
* Cervical radiculopathy, thoracic outlet syndrome,
* Malignant condition,
* Have systemic diseases such as neurological, psychological, cardiovascular, rheumatology and loss of function due to these diseases,
* Previous surgery history in the spine and upper extremity, including the cervical and lumbar region,
* Fracture in the spine and upper extremity, including the cervical and lumbar region, with an inflammatory history,
* Acute infection,
* Continuing another rehabilitation program,
* Individuals who do not agree to participate in the study and do not give written consent will be excluded from the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2021-04-14 (Actual); Primary Completion 2023-02-20 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
Evaluation of Muscle Thickness with Ultrasonography | 15 minutes, through study completion, an average of 8 weeks, Change from Baseline Muscle Thickness at 8 weeks
  Ultrasonography is used to evaluate the architectural properties of the muscle (such as thickness) in chronic painful musculoskeletal problems such as neck-back pain. Muscle architecture measurements with ultrasound will be carried out before and after the exercise program by the specialist radiology doctor who is blind to the results of the study using 3.5-10 MHz convex and linear probes (Soundcam Mobile Ultrasound Device). Within the scope of our study, the muscle thickness of the spinal muscles will be evaluated in the resting position.
Evaluation of Functional Capacity Level with Functional Capacity Assessment Test | 20 minutes, through study completion, an average of 8 weeks, Change from Baseline Functional Capacity Level at 8 weeks
  Functional capacity assessment evaluates the effectiveness (time to completion, weight it can handle) of each activity that includes different activities for neck pain. The test includes the activities of "repetitive reaching out, lifting objects overhead, working overhead". The validity and reliability of the Functional Capacity Assessment Test in individuals with chronic neck pain has been shown. The time individuals can complete the tests will be recorded.
Evaluation of Functional Capacity Level with Back Performance Scale | 10 minutes, through study completion, an average of 8 weeks, Change from Baseline Functional Capacity Level at 8 weeks
  The back performance test (Back Performance Scale) is a test that evaluates the effectiveness of each activity that includes 5 different activities (socks test, gathering test, righting test, fingertip-floor test, carrying test). The Back Performance Scale test is scored between 0-15 points. An increase in score indicates a poor result.

SECONDARY OUTCOMES:
Evaluation of quality of life | 5 minutes, through study completion, an average of 8 weeks, Change from Baseline quality of life at 8 weeks
  Quality of life Assessment: SF-36 SF-36 is a scale consisting of 36 questions that evaluates the health status of the person with 8 sub-items (physical function, role limitations, social function, mental health, vitality, pain, general health). Scoring between 0-100 is made separately for each sub-item. It indicates good health as the score approaches 100. The validity and reliability study, Koçyiğit et al. Made by.
Evaluation of Exercise Adaptation Assessment: Exercise Adaptation Rating Scale (EUAS) | 5 minutes, through study completion, an average of 8 weeks, Change from Baseline Exercise Adaptation Assessment at 8 weeks
  It will be evaluated using the Exercise Adherence Rating Scale (EARS), which evaluates exercise compliance (52). The first 2 parts of the scale consist of 6 questions and the third part consists of 10 questions. The first part is not included in the scoring and the maximum score to be obtained from two parts is 64. An increase in score indicates an increased adaptation to exercise. The Turkish validity and reliability study of the scale was conducted in 2019 by Korkmaz et al.
Evaluation of Difficulty of Functional Activities and Exercise Program Satisfaction (GAS) | 5 minutes, through study completion, an average of 8 weeks, Change from Baseline Difficulty of Functional Activities and Exercise Program Satisfaction at 8 weeks
  VAS is used in measurement by digitizing the values that cannot be measured numerically. It is a line measurement, often on a 10 cm long horizontal or vertical line, where the person indicates his condition. Pain is used in the literature to evaluate satisfaction. In the satisfaction evaluation, it is evaluated as "0: there was no decrease in complaints, I am not satisfied, 10: complaints completely disappeared, I am very satisfied". In the study, the functional activity difficulty will be evaluated as "0: Being unable to do the activity, 10: Being able to do the activity at the level before the neck pain started".

CONTACTS AND LOCATIONS:
Locations (1):
- Yasemin Özel Aslıyüce, Ankara, Sıhhiye, Turkey (Türkiye)